CLINICAL TRIAL: NCT00932256
Title: STAHIST IND 105781 Phase 1 Clinical Trial
Brief Title: Clinical Trial of STAHIST in Seasonal Allergic Rhinitis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Magna Pharmaceuticals, Inc. (Industry)
Responsible Party: Warren P. Lesser, President, MAGNA Pharmaceuticals, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STAHIST IND 105781; NCT00931658 (obsolete NCT alias)
Record Dates: First submitted 2009-06-30; First posted 2009-07-03 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-12

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Rhinitis, Allergic, Seasonal
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- STAHIST for seasonal allergic rhinitis (Experimental): STAHIST for seasonal allergic rhinitis: each white, scored tablet contains pseudoephedrine hydrochloride 90mg, chlorpheniramine maleate 8mg, and atropine sulfate .24mg
  Interventions: Drug: STAHIST NDC #58407-536-01

INTERVENTIONS:
Drug: STAHIST NDC #58407-536-01 — Oral tablet containing Pseudoephedrine hydrochloride 90mg, chlorpheniramine maleate 8mg, atropine sulfate .24mg, one tablet BID.
  Other Names: STAHIST NDC#58407-536-01

SUMMARY:
MAGNA intends to show that the combination of pseudoephedrine, chlorpheniramine, plus a small amount of belladonna alkaloid is a comprehensive, safe and effective twice daily (BID) drug treatment for seasonal allergic rhinitis (SAR) patients with post-nasal drip (PND). The phase 1 single-dose trial will consist of 21 subjects: 1) to gather pharmacodynamic measurements and blood levels of active ingredients over 12 hours; 2) To report subjective scores by subjects rating efficacy of single dose of STAHIST; 3) To report any side effects or adverse drug reactions and rate the severity of incidence.

DETAILED DESCRIPTION:
No procedure will be performed until Informed Consent has been obtained. Inclusion and exclusion criteria will be verified. Subjects will be required to stop using oral nasal decongestants or first generation antihistamines for 48 hours, second generation antihistamines and Singulair for seven days, systemic corticosteroids for 30 days, and nasal or ocular corticosteroid medications for two weeks. Use of these drugs will not be allowed during the study.

Blood samples will be drawn at specific time points: baseline fasting blood draw just before 7AM, then at 9 AM, 11AM, 3PM, and 7PM. A single oral dose of STAHIST will be administered at 7AM.

During the study a diary of the five study symptoms (S5 Diary) will be scored hourly over the 12-hour period as follows: 0 none, 1 mild, 2 moderate, 3 severe. The S5 symptoms are 1. Nasal Congestion (Stuffiness); 2. Sneezing; 3. Rhinorrhea (runny nose); 4. Nasal Itching; 5. Post-nasal drip. Post nasal drip is defined for the patient as "you can feel accumulated mucus dripping down the back of your throat from your sinuses, also possibly including a tickly cough or sore throat due to this sensation of mucus."

Side effects or adverse drug reactions will be scored if they occur and hourly as 1 mild, 2 moderate, and 3 severe. Any adverse events will be recorded. Any subject who is not able or who is unwilling to continue keeping a diary or participate in blood draws will be permitted to withdraw from the study. Safety will be assured by the frequent visible assessment and questioning of subjects as well as monitoring of subjects' vital signs by Dr. Pollard and his nursing staff. Subjects will remain in the clinic during the 12-hour dosage interval. Thereafter, Dr. Pollard and selected staff will be on call 24 hours to answer any subject phone calls.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of any ethnic group between the ages of 18 and 60 years of age.
* History of moderate to severe SAR for at least one year.
* Subjects' symptoms will include the five symptoms ("S5") that are the focus of this study:

  * nasal congestion;
  * rhinorrhea;
  * nasal itching;
  * sneezing;
  * post nasal drip.
* Prior to study subjects' good health will be confirmed by medical history and physical examination.
* Allergic hypersensitivity will be confirmed by an appropriate test as deemed necessary by the physician or well established medical history.

Exclusion Criteria:

* Pregnancy or lactation.
* Immunotherapy unless at stable maintenance dose.
* Presence of a medical condition that might interfere with treatment evaluation or require a change in therapy including but not limited to high blood pressure or urinary retention problems.
* Alcohol dependence.
* Use of any other investigational drug in the previous month.
* Subjects presenting with asthma requiring corticosteroid treatment.
* Subjects with multiple drug allergies.
* Subjects known to have an idiosyncratic reaction to any of the ingredients in STAHIST.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2009-10; Primary Completion 2009-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To gather pharmacodynamic measurements and assess blood levels (five draws) of the active ingredients in STAHIST over the dosage interval period of 12 hours. | August 2009

SECONDARY OUTCOMES:
To report any side effects or adverse drug reactions and rate the severity of incidence. | August 2009

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Pollard, MD, Principal Investigator — Family Allergy and Asthma Research Institute
Locations (1):
- Family Allergy and Asthma Research Institute, Louisville, Kentucky, United States

REFERENCES:
- [Result] Moffitt EM. Symptomatic management of upper respiratory allergies. J Miss State Med Assoc. 1968 Apr;9(4):159-61. No abstract available. PMID 5640510